CLINICAL TRIAL: NCT05063006
Title: Exercise Tolerance in Patients With Implanted Left Ventricular Assist Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karol Wierzbicki (Other)
Collaborators: Cor Aegrum Foundation of Cardiac Surgery Development in Cracow, Poland (Unknown); Medtronic Poland Spółka z ograniczoną odpowiedzialnością (Industry); AGH University of Science and Technology, Krakow, Poland (Unknown)
Responsible Party: Sponsor-Investigator, Karol Wierzbicki, Head of Cardiac Transplantation and Mechanical Circulatory Support Unit, John Paul II Hospital, Krakow
Organization: John Paul II Hospital, Krakow (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: NB.0710.003.2021P
Record Dates: First submitted 2021-09-16; First posted 2021-09-30 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Left Ventricular Assist Device
Keywords: left ventricular assist device; cardiopulmonary exercise test; stress echocardiography; heart failure; mechanical circulatory support; peak VO2
MeSH Terms: conditions — Heart Failure | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: prospective crossover AB/BA study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LVAD pump speed dynamically adjusted (Experimental)
  Interventions: Other: Cardiopulmonary exercise test with gradually increased pump speed depending on live echocardiographic imaging.
- LVAD pump at optimal resting speed (Active Comparator)
  Interventions: Other: Cardiopulmonary exercise tests with maintained baseline optimal pump speed settings.

INTERVENTIONS:
Other: Cardiopulmonary exercise tests with maintained baseline optimal pump speed settings. — Optimal resting LVAD speed settings is defined as periodic aortic valve opening while maintaining the central position of the intraventricular septum, minimizing mitral regurgitation, and preserving the mean systemic blood pressure above 65 mmHg. The aim is to achieve an aortic valve opening ratio of around 25-33% by changing the pump speed at resting conditions.
  Arms: LVAD pump at optimal resting speed
Other: Cardiopulmonary exercise test with gradually increased pump speed depending on live echocardiographic imaging. — During the modified speed exercise, when the aortic valve opening ratio rises above 50%, the pump speed is increased by 100 revolutions per minute (RPM). As the aortic valve remains closed the RPM is lowered by 100. Speed increment is not greater than 100 RPM per 45 seconds to enable an echocardiographic analysis of resulting changes and prevent suction events. There is no determined target speed, neither per time period nor maximal.
  Arms: LVAD pump speed dynamically adjusted

SUMMARY:
To evaluate the concept of dynamic pump speed optimization based on the echocardiographic assessment of aortic valve opening during cardiopulmonary exercise test.

DETAILED DESCRIPTION:
Left ventricular assist devices (LVAD) are becoming a destination therapy in patients with end-stage left ventricular dysfunction. Current generation pumps operate with a fixed rotation speed without the capability of automated speed adjustment. It was shown that acceleration of the pump speed during stress test increases the maximum exercise tolerance. Periodic aortic valve opening (AVO) is used to set up an optimal resting pump speed. The study aimed to evaluate the concept of dynamic pump speed optimization based on the echocardiographic assessment of AVO during the cardiopulmonary exercise test (CPET).

Patients with implanted third-generation LVADs with hydrodynamic bearing (HVAD, Medtronic, MN, USA) are prospectively enrolled. Two CPETs are performed after resting speed optimization. The first one with maintained baseline pump speed settings, and the second one with gradually increased speed depending on live echocardiographic imaging. The sequence of tests is random.

ELIGIBILITY:
Inclusion Criteria:

* Patients with implanted cardioverter-defibrillator and third-generation centrifugal CF-LVAD with hydrodynamic bearing (HVAD, Medtronic, Minnesota, United States), at least three months after surgery.

Exclusion Criteria:

* Hemodynamic instability.
* Non-therapeutic anticoagulation.
* Device or intracardiac thrombus.
* Inflammation.
* Active bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-08-04 (Actual)

PRIMARY OUTCOMES:
Echocardiographic appraisal of aortic valve opening during cycle ergometer exercise. | Immediately, during cycle ergometer exercise
  Assessment of aortic valve opening during cycle ergometer exercise in LVAD patients.

SECONDARY OUTCOMES:
Change in oxygen consumption | Immediately, during cycle ergometer exercise
  By using the cardiopulmonary exercise test
Change in perceived exertion | Immediately, during cycle ergometer exercise
  By using the Borg rating of perceived exertion scale. Score 6-20 (6 - no exertion, 20 - maximal exertion)
Change in pump speed | Immediately, during cycle ergometer exercise.
  By assessing pump speed (RPM)
Change in pump flow | Immediately, during cycle ergometer exercise
  By assessing pump flow (l/min)
Change in pump power | Immediately, during cycle ergometer exercise
  By assessing pump power (W)

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Stapor, MD PhD, Study Director — Department of Interventional Cardiology, John Paul II Hospital; Karol Wierzbicki, Assoc Prof, Principal Investigator — Department of Cardiovascular Surgery and Transplantology, John Paul II Hospital
Locations (1):
- John Paul II Hospital, Krakow, Lesser Poland Voivodeship, Poland